CLINICAL TRIAL: NCT04478526
Title: Determining the Efficacy of Online Cognitive Behavioural Therapy for Generalized Anxiety Disorder Compared to Pharmaceutical Interventions
Brief Title: Efficacy of Online CBT for GAD Compared to Pharmaceutical Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Nazanin Alavi (Other)
Collaborators: Online PsychoTherapy Clinic (Other)
Responsible Party: Sponsor-Investigator, Dr. Nazanin Alavi, Principal Investigator, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSIY-604-18
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; Online Psychotherapy; Cognitive Behavioural Therapy
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Selective Serotonin Reuptake Inhibitors; Serotonin and Noradrenaline Reuptake Inhibitors; Serotonin

STUDY DESIGN:
Intervention Model Description: This study has been designed using a quasi-experimental design to allow patients the freedom to choose which treatment modality they would like to participate in. This research design aims to be naturalistic by mimicking the decisions made by patients and physicians regarding the course of treatment and type of pharmacotherapy prescribed within mental health services across Ontario. The treatments provided within the study also aim to replicate evidence-based best practice clinical guidelines for the treatment of GAD. Arms include eCBT, eCBT + Pharmacotherapy, Pharmacotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- e-CBT (Experimental): Weekly sessions of e-CBT through OPTT will consist of approximately 30 slides. Each session is expected to last approximately 50 minutes. The content and format of each weekly online session were designed to mirror live CBT. The slides will highlight a different topic each week and include general information, an overview of skills and homework on that topic. The homework included in each session will be submitted through OPTT and reviewed by the clinicians with personalized feedback provided by clinicians within three days of submission. Weekly homework submission for feedback will be mandatory before being eligible for the next session. Biweekly GAD-7, DASS-42 and Q-LES-SF questionnaires will be completed through OPTT. A second STAI will be completed in the final week of e-CBT treatment.
  Interventions: Behavioral: Electronic Cognitive Behavioural Therapy
- Pharmacotherapy (Experimental): Biweekly meeting with psychiatrist with GAD-7, DASS-42 and Q-LES-SF. Pharmacotherapy class decided according to protocol developed in accordance with Canada's best practice guidelines for GAD treatment. At second appointment, medication will be maintained and optimized, regardless of response. At third appointment, optimized if partial response or switched according to protocol if no response. Partial response is improvement of 20% or more in GAD-7. If switched, 6-week protocol will recommence with new medication. At fourth appointment, dosage optimized if responding well to medication and improvement greater than 50% within primary arm, or 20% if secondary arm, patient will remain on said medication for remainder of 12-week study. If not improving more than 20%, medication switched according to protocol and 6-week protocol will recommence. If primary arm and 20-50% improvement after six weeks on new medication, augmented with olanzapine, risperidone or benzodiazepines.
  Interventions: Drug: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors)
- e-CBT + Pharmacotherapy (Experimental): Participants will commence both treatments described above simultaneously.
  Interventions: Drug: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors); Behavioral: Electronic Cognitive Behavioural Therapy

INTERVENTIONS:
Drug: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors) — If never taken SSRI or SNRI, commence primary medication arm (SSRI: sertraline, escitalopram or Pregabalin/SNRI: duloxetine, venlafaxine) will be described to patient and will begin either. If deemed unresponsive to either prior to study, commence medication they have not been previously unresponsive to. Unresponsive if GAD did not improve after treatment with maximum tolerated dose for 8-weeks. If deemed unresponsive to SSRI and SNRI/pregabalin, commence secondary medication arm (bupropion/mirtazepine, buspirone/imipramine) with both being described to patient and begin either. Switch protocol: If unresponsive after 4 or 6 weeks, switch to another class. If started in primary or secondary and not previously demonstrated non-response to second class of medications within arm, switch to second class within arm. If started in primary and previously deemed unresponsive to second class, begin secondary if non-response indicates switch necessary.
  Arms: Pharmacotherapy; e-CBT + Pharmacotherapy
Behavioral: Electronic Cognitive Behavioural Therapy — Weekly sessions of e-CBT through OPTT will consist of approximately 30 slides. Each session is expected to last approximately 50 minutes. The content and format of each weekly online session was designed to mirror live CBT. The slides will highlight a different topic each week and include general information, an overview of skills and homework on that topic. The homework included in each session will be submitted through OPTT and reviewed by the clinicians with personalized feedback provided by clinicians within three days of submission. Weekly homework submission for feedback will be mandatory before being eligible for the next session. Biweekly GAD-7, DASS-42 and Q-LES-SF questionnaires will be completed through OPTT. A second STAI will be completed in the final week of e-CBT treatment.
  Arms: e-CBT; e-CBT + Pharmacotherapy

SUMMARY:
Generalized anxiety disorder (GAD) is an extremely prevalent and debilitating mental health disorder. Currently, the gold standard treatment for GAD is cognitive behavioural therapy (CBT) and/or pharmacotherapy. The most common medications used to treat GAD are selective serotonin reuptake inhibitors (SSRIs) and selective norepinephrine reuptake inhibitors (SNRIs). While CBT is a gold standard treatment for GAD, it is costly, time-consuming, and often inaccessible. Fortunately, the electronic delivery of CBT (e-CBT) has emerged as a promising solution to address these barriers. e-CBT has shown to offer comparable results to in-person CBT while improving accessibility for patients and time efficiency for clinicians. The following project aims to investigate the treatment efficacy of e-CBT compared to, and in conjunction with pharmacotherapy for GAD. This study has been designed using a quasi-experimental design to allow patients the freedom to choose which treatment modality they would like to receive. Participants with a diagnosis of GAD will be enrolled in 1 of 3 possible treatment arms: e-CBT, medication, or combination. The e-CBT program will include a 12-week psychotherapy program delivered through the Online Psychotherapy Tool (OPTT), a secure, cloud-based, digital mental health platform. The treatment efficacy of e-CBT will be compared to the treatment efficacy of the medication arm and the combination arm. Conclusions: If e-CBT is shown to either be comparable to medication or that the effects of both treatments are augmented when used in tandem, these findings could have major implications on the mental health care system. e-CBT is a more accessible, and affordable treatment that could increase mental health care capacity by four-folds if proven viable.

DETAILED DESCRIPTION:
Methodology Research Design. This study has been designed using a quasi-experimental design to allow patients the freedom to choose which treatment modality they would like to participate in. This research design aims to be naturalistic by mimicking the decisions made by patients and physicians regarding course of treatment and type of pharmacotherapy prescribed within mental health services across Ontario. The treatments provided within the study also aim to replicate evidence-based best practice clinical guidelines for treatment of GAD.

Research Participants. Patients will be referred to the study by primary care physicians within Toronto and Kingston, Ontario. Patients will be referred to the Anxiety Outpatient Clinic at the Hotel Dieu Hospital site of Kingston Health Sciences Centre or the Mood and Anxiety Clinic within the Centre for Addiction and Mental Health (both sites herein referred to as "the clinic"). Upon receiving a referral to the clinic, participants will be contacted by the study's Research Coordinator and asked to indicate their interest (or lack thereof) in the study. If interest is indicated and the study's inclusion criteria are met, the patient will have a study intake appointment scheduled for the same day as their intake appointment at the clinic. To be considered for inclusion within the study, patients must:

* be 18 years of age or older
* have consistent and reliable access to the internet
* be diagnosed with GAD according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) by a clinician
* meet the criteria for GAD according to the GAD-7 Screener (GAD-7)
* Be competent to consent to participate
* Speak and read English Patients will be deemed ineligible for participation in the study if they are in acute distress.

Allocation of Subjects between Arms of the Study. Subjects will be presented with all three arms of the study within their study intake appointment by the Research Coordinator. After obtaining informed consent, patients will meet with one of the study's psychiatrists during their clinic intake appointment and discuss the recommended treatment plan. In collaboration with the psychiatrist, patients will decide whether or not they would like to begin pharmacotherapy and/or e-CBT treatment.

Criteria for Discontinuation. Patients' participation in the study will be discontinued if they are found to be noncompliant to their treatment. This will be defined as stopping medications all together or reportedly skipping more than two days in a row of medication. Patients will be found noncompliant with e-CBT treatment if they miss more than two weeks of e-CBT sessions or fail to complete weekly homework assignments. Patients' participation within the study will also be halted if they are deemed to be in acute crisis by self-report or the psychiatrist in charge of their care.

Study Protocol. After being referred to the study by a clinician uninvolved within the study, patients will be contacted by the Research Coordinator to determine the patient's interest in participating in the study. If interest is indicated, an intake appointment for the study will be scheduled for the same date as the intake appointment to the clinic.

Intake appointment. Upon attending the intake appointment, the Research Coordinator will explain all three arms of the study and review the study's letter of information. After sufficient time has been provided to ensure the patient understands the study, informed consent will be obtained by the Research Coordinator and the patient will complete the State Trait Anxiety Inventory (STAI), a demographics questionnaire, Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-QSF), GAD-7 and the 42-item Depression Anxiety Stress Scales (DASS-42). Following the intake appointment, patients will, in collaboration with their psychiatrist, decide on which treatment modalities they would like to participate in (e-CBT and/or pharmacotherapy). Treatment will then proceed according to the arms below, with patients participating in e-CBT and pharmacotherapy commencing both arms simultaneously within their clinic intake appointment.

e-CBT. Weekly sessions of e-CBT through OPTT will consist of approximately 30 slides. Each session is expected to last approximately 50 minutes. The content and format of each weekly online session was designed to mirror live CBT. The slides will highlight a different topic each week and include general information, an overview of skills and homework on that topic. The homework included in each session will be submitted through OPTT and reviewed by the clinicians with personalized feedback provided by clinicians within three days of submission. Weekly homework submission for feedback will be mandatory before being eligible for the next session. Biweekly GAD-7, DASS-42 and Q-LES-SF questionnaires will be completed through OPTT. A second STAI will be completed in the final week of e-CBT treatment.

Pharmacotherapy. If patients chose to participate in the pharmacotherapy stream of treatment, they will attend biweekly medication reconciliation appointments with their psychiatrist at the clinic. If the patient is participating solely in the pharmacotherapy arm, they will complete the biweekly GAD-7, DASS-42 and Q-LES-SF within each of their appointments. If the patient is completing both pharmacotherapy and e-CBT, questionnaires will only be completed through OPTT. Upon attending their clinic intake appointment, the patient's medication history (including any current medications) will be collected and all medications prescribed for GAD prior to the study will be switched to the medications suggested in the protocol and if needed to be continued the dose will be unchanged 6 weeks prior to start of the study and during the study. Within the patient's clinic intake appointment, they will commence pharmacotherapy with the medication class decided according the "starting medication" protocol below, which was developed in accordance with Canada's best practice guidelines for the treatment of GAD. The pharmacotherapy protocol is summarized in Figure 1.

General 6-week protocol. At the patient's second appointment (2 weeks on the medication), their medication will be maintained and optimized, regardless of whether or not a response is reported. At the patient's third appointment (4 weeks on the medication), the medication will be optimized if a partial response is reported or the medication will be switched according to the "medication switch protocol" if no response is reported. Partial response will be defined as an improvement of 20% or greater in their GAD-7 score compared to baseline. If the medication is switched (the patient reports less than a 20% improvement in their GAD-7 score compared to baseline), the 6-week protocol will recommence with the new medication. At the patient's fourth appointment (6 weeks on the medication), their dosage will be optimized if the patient is responding well to the medication and reports an improvement greater than 50% if within the primary medication arm, or 20% if within the secondary medication arm, in their GAD-7 score compared to baseline, the patient will remain on said medication for the remainder of the 12-week study. If the patient does not report an improvement of more than 20% in their GAD-7 score compared to baseline, the patient's medication will be switched according to the "medication switch protocol" and the 6-week protocol will recommence with the new medication. If the patient is within the primary medication arm and reports a 20-50% improvement in GAD symptoms compared to baseline after six weeks on the new medication, the medication with be augmented with either olanzapine, risperidone or benzodiazepines.

Starting Medication. If the patient has never taken an SSRI or SNRI, the patient will commence the primary medication arm. The two classes of medications within the primary arm will be described to the patient and, with the recommendation of the prescribing psychiatrist, the patient will begin either an SSRI (sertraline or escitalopram) or pregabalin/an SNRI (duloxetine or venlafaxine).

If, prior to the beginning of the study, the patient has been deemed unresponsive to either an SSRI or an SNRI/pregabalin, the patient will commence the primary medication arm. The patient will start the medication class that they have not been previously deemed unresponsive to (i.e., if previously unresponsive to sertraline, the patient will commence the SNRI class). A patient will be considered previously unresponsive if their anxiety did not improve after treatment with the maximum tolerated dose of the specific medication for an eight-week duration.

If the patient has been deemed unresponsive to both an SSRI and an SNRI/pregabalin, the patient will commence the secondary medication arm. The two classes of medications within the secondary arm will be described to the patient and, with the recommendation of the prescribing psychiatrist, the patient will begin either bupropion/mirtazepine or buspirone/imipramine.

Medication switch protocol. If the patient is deemed unresponsive to a medication after 4 or 6 weeks of administration (the patient reports less than a 20% improvement in their GAD-7 score compared to baseline), their medication should be switched to another class. If the patient has a history of non-response to any of the four medication classes, these classes should be removed as pharmacotherapy options for their treatment within the study (i.e., if a patient was deemed unresponsive to SSRIs prior to commencing the study, the patient should not be prescribed sertraline or escitalopram at any point within the study). If the patient was started in the primary or secondary medication arm and has not previously demonstrated non-response to the second class of medications within that arm, the patient should be switched to the second class of pharmaceuticals within that arm. If the patient was started in the primary arm and was previously deemed unresponsive to the second class of pharmaceuticals within that arm, the patient should begin the secondary medication arm if non-response indicates a medication switch is necessary.

Six Month Follow-up. All patients will be contacted through telephone by the Research Coordinator 6 months after their 12 weeks within the study have ended to complete follow-up questionnaires. The patients will complete a third STAI and another Q-LES-SF, DASS-42 and GAD-7. These measurements will act to determine the longevity of treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have consistent and reliable access to the internet
* Be diagnosed with GAD according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) by a clinician
* Meet the criteria for GAD according to the GAD-7 Screener (GAD-7)
* Be competent to consent to participate
* Speak and read English

Exclusion Criteria:

- Patients will be deemed ineligible for participation in the study if they are in acute distress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Change in State Trait Anxiety Level | Baseline, week 2, 4, 6, 8, 10, 12, plus 6-month follow-up
  State Trait Anxiety Inventory (STAI) - Scale: 1-4 (1 = not at all, 4 = very much)
Change in Quality of Life | Baseline, week 2, 4, 6, 8, 10, 12, plus 6-month follow-up
  Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-QSF) - Scale: 1-5 (1 = very poor, 5 = very good)
Change in Generalized Anxiety Levels | Baseline, week 2, 4, 6, 8, 10, 12, plus 6-month follow-up
  Generalized Anxiety Disorder - 7 (GAD-7) - Scale: 0-3 (0 = never, 3 = nearly every day)
Change in Depression and Anxiety Scale | Baseline, week 2, 4, 6, 8, 10, 12, plus 6-month follow-up
  42-item Depression Anxiety Stress Scales (DASS-42) Scale: 0-3 (0 = not at all, 3 = very much)

SECONDARY OUTCOMES:
Demographics Information | Baseline, week 2, 4, 6, 8, 10, 12, plus 6-month follow-up
  Demographic questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Alavi, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Information from study is confidential and anonymity will be protected. Each patient participating in e-CBT will have password-protected encrypted file through web-based platform OPTT. Questionnaires and homework submitted via OPTT can only be accessed by psychiatrists involved within study and participating clinicians. Data from research will be saved without mention of patient names with all patients being identified with unique identification number in all data from this study. Master file of participant ID numbers and participant names will be maintained in password-protected encrypted file and destroyed once study has been completed. Hard copies files will be stored in locked cabinets and offices and will be available only to clinicians providing treatment and Research Coordinator. Participants will not be identified in any publication or reports and electronic data will be saved in password-protected encrypted files for 5 years after last publication then permanently destroyed.

REFERENCES:
- [Derived] Alavi N, Stephenson C, Yang M, Shirazi A, Shao Y, Kumar A, Yee CS, Miller S, Stefatos A, Gholamzadehmir M, Abbaspour Z, Patel A, Patel C, Reshetukha T, Omrani M, Groll D. Determining the Efficacy of Electronic Cognitive Behavioral Therapy for Generalized Anxiety Disorder Compared to Pharmaceutical Interventions: Protocol for a Quasi-Experimental Study. JMIR Res Protoc. 2021 May 27;10(5):e27772. doi: 10.2196/27772. PMID 33857917
- See also: Publication — https://www.frontiersin.org/journals/psychiatry/articles/10.3389/fpsyt.2023.1194955/full